CLINICAL TRIAL: NCT04417296
Title: IMPACTS OF BRAXTON-HICKS CONTRACTIONS ON COMPUTERISED CARDIOTOCOGRAPHY PARAMETERS: A POTENTIAL LINK.
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Marco La Verde, MD, research , gynecology and obstetrics, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 004
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Braxton Hicks' Contractions
Keywords: Braxton Hicks' contractions; uterine contractions; fetal well-being; Computerized cardiotocography (cCTG); Fetal heart rate (FHR); Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nonlaboring term singleton pregnancies: All patients had an uncomplicated pregnancy and to define a pregnancy uncomplicated we adopted Chappell's definition: "a normotensive pregnancy, delivered at >37 weeks, ending in a live-born baby who was not small for gestational age and did not have any other notable pregnancy complications"
  Interventions: Diagnostic Test: antepartum computerised cardiotocography analysis

INTERVENTIONS:
Diagnostic Test: antepartum computerised cardiotocography analysis — A common obstetric methodical to evaluate the fetal well-being is the antepartum fetal heart rate (FHR) monitoring through cardiotocography (CTG)

SUMMARY:
Several types of research examined the relationship of Braxton-Hicks contractions and uterine flow. Nevertheless, no one considered the relationship of the maternal perception of Braxton-Hicks contractions with the fetal wellbeing quantifies through computerised cardiotocography. Our study wants to estimate the correlation between the maternal perception of Braxton-Hicks contractions and antepartum computerised cardiotocography parameters.

ELIGIBILITY:
Inclusion Criteria:

* Nonlaboring women with a term uncomplicated singleton pregnancy

Exclusion Criteria:

* complicated singleton pregnancy

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We included pregnant who were referred for the fetal antepartum cardiotocography monitoring to the outpatient clinic of the "Luigi Vanvitelli" University of Campania in Naples, Italy. All patients had an uncomplicated pregnancy and to define a pregnancy uncomplicated we adopted Chappell's definition: "a normotensive pregnancy, delivered at >37 weeks, ending in a live-born baby who was not small for gestational age and did not have any other notable pregnancy complications"
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
the comparison of the antepartum computerised cardiotocography between the patients with Braxton-Hicks contractions and the patients without uterine activity | pre-intervention
  External cCTG was completed at least 20 minutes (maximum 60 minutes), two transducers were placed on the maternal abdomen: one over the fetal heart level and the other one at the uterine fundus. For each cCTG, the following data were evaluated: Basal FHR

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli studi della Campania "Luigi Vanvitelli"- OB & Gyn -, Napoli, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided